CLINICAL TRIAL: NCT03341611
Title: A Neuroeconomic Study of Choice Consistency in Aging
Brief Title: The Effect of Aging on Value Based Decision-making
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Isabelle Brocas, Professor of Economics, University of Southern California
Other Study IDs: 1R21AG046917-01A1 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Healthy Aging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults 55 and younger
  Interventions: Behavioral: Neuro-imaging during behavioral decision-making task
- Adults 55 and older
  Interventions: Behavioral: Neuro-imaging during behavioral decision-making task

INTERVENTIONS:
Behavioral: Neuro-imaging during behavioral decision-making task — All participants will make simple decisions while in a scanner.

SUMMARY:
The investigators propose to study the effect of aging on the neural circuitry involved in valuation and value reasoning and to relate it to choice anomalies and inconsistencies. Quantifying and characterizing valuation-based decision-making deficits in older adults, and their relationship to the aging brain, can inform and facilitate intervention - both at the level of the individual and at the level of policy.

DETAILED DESCRIPTION:
The attribution of value to prospects is a fundamental element of decision-making, as most day-to-day decisions involve comparing items. Studies on aging document behaviors reflecting difficulties in making comparisons between options, in particular when those options are complex. Given the growing complexity of economic products (insurance, savings, mortgages or even telephone plans), older adults may have difficulty making decisions that accurately reflect their underlying preferences. It is plausible that this difficulty is linked to age-related brain function decline within sectors of the lateral prefrontal cortex implicated in working memory and cognitive control. This study assesses age-related changes in how the brain computes value and makes value comparisons using a well-established economic paradigm, the "generalized axiom of revealed preference" (GARP) Task, that tests the internal consistency of a subject's preferences by offering repeated choices between bundles of goods. A preliminary study suggests that aging is associated with greater GARP-Task inconsistency. Although the neural correlates of GARP inconsistency have not been directly established, indirect evidence suggests that the medial orbitofrontal cortex is important in all value-based decision-making, and that areas in the lateral prefrontal and parietal cortices (fronto-parietal network) are important for maintaining consistency in complex decisions (e.g., multi-attribute decisions). Aging is associated with structural and functional deficits within the fronto-parietal network. Therefore, the investigators believe that studying the neural correlates of the GARP-Task is a promising approach to investigate decision-making deficits in aging. The investigators will recruit 45 young adults, and 45 old adults. Participants will complete the GARP-Task and an functional Magnetic resonance imaging (fMRI) variant designed to isolate neural correlates of valuation of single items, of multiple instances of the same item ("scaling") and of sets of distinct items ("bundles"). Brain activity will be related to diagnosis and to variance in GARP-Task inconsistency. Given the prominence of age-related decline in working memory, the investigators hypothesize that age will be associated with higher GARP-Task inconsistency and to deficits in conditions that require manipulation of value signals (scaling and bundles). The investigators anticipate that these deficits will be associated with low recruitment within the fronto-parietal network and with reduced functional connectivity between this network and the medial Orbitofrontal Cortex (OFC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* 1- Subjects under 18yo . 2- Subjects with known cognitive disorders 3- Subjects with visual or auditory deficits that would interfere with the ability to complete the experimental tasks.

  4- Subjects reporting having metal implants 5- Subjects with a history of major anxiety disorder or other major psychiatric condition, 6- Subjects with a documented or subjectively reported claustrophobia. 7- Subjects thinking they are or may be pregnant. 8- Subjects with a history of head trauma that resulted in loss of consciousness for more than 5 minutes.

  9-Hx of seizures 10-Left Handed 11- On any medications affecting cognition 12- For tasks involving foods: a) Currently on diet and or b) any known food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults above 18yo
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Computerized behavioral choice task | 2 hours
  The task consists in 450 trials. In each trial, the participant needs to choose between food items presented on a computer screen. Frequency of choices is used to assess the ranking (or value) of these food items and inconsistencies in choices are recorded. Food items vary in complexity (from single items to complex bundles).
Brain imaging to track brain regions involving in value | 1 hour
  fMRI images are collected during part of the behavioral choice task. Behavioral measures are used to track value encoding as well as inconsistent choices in the brain (as a function of item complexity). These data are eventually aggregated across participants in each condition (using standard methods) to identify the regions of interest involved in our experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Brocas, PhD, Principal Investigator — University of Southern California
Locations (1):
- LABEL, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all data and results.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
URL: http://dornsife.usc.edu/label/